CLINICAL TRIAL: NCT00746148
Title: Reflexology's Effect on Polycystic Ovary Syndrome (REPOS): A Pilot Study
Brief Title: Reflexology's Effect on Polycystic Ovary Syndrome: A Pilot Study
Acronym: REPOS
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: dmw1
Record Dates: First submitted 2008-09-02; First posted 2008-09-03 (Estimated); Last update posted 2012-12-04 (Estimated); Status verified 2012-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Reflexology; Complementary and Alternative Medicine; Endocrinopathy; Oligo; Amenorrhoea
MeSH Terms: conditions — Polycystic Ovary Syndrome; Endocrine System Diseases; Amenorrhea | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Reflexology
  Interventions: Other: Reflexology
- 2 (No Intervention): No intervention

INTERVENTIONS:
Other: Reflexology — 10 weekly sessions of 45 minutes each
  Arms: 1

SUMMARY:
Polycystic Ovary Syndrome (PCOS) is very common, affecting approximately 5% of women of reproductive age, and impacts not only on quality of life, but also has long-term health consequences for many sufferers, such as increased risks of developing Type II diabetes, cardiovascular disease and cancer of the womb. The symptoms that may occur such as irregular periods; lots of body hair; thinning hair on scalp, obesity and infertility, can also lead to poor self-esteem. Whilst treatments can help fertility, other treatments to correct the other symptoms are less successful. Alternative methods to regulate periods would be helpful, especially ones which avoid the long-term use of steroids in patients who may already be overweight. Reflexology is poorly represented in scientific papers, with nothing published regarding reflexology and its effect upon PCOS. However patients who use reflexology report more regular periods, thicker hair on scalp and greater wellbeing. Therefore we aim to investigate the effect of reflexology on:

1. The menstruation cycle (normal being every 21-35 days).
2. Imbalances in hormone, insulin and blood sugar levels associated with PCOS.
3. Other problems associated with PCOS such as thinning hair on scalp, excessive body hair, and obesity.
4. Quality of life. Government and NHS agendas agree that if there's evidence of an effective complimentary therapy the NHS should provide it. Therefore the results may have an influence on the care pathways of patients with PCOS towards a more holistic, patient centred and empowered approach. It is also non invasive and liable to result in higher patient satisfaction regarding their treatment. This research may also inform policy makers so that complementary medicine provision is provided on a wider basis within the NHS, which at the moment is dictated by the individual Trust's budget allocation. However this research could save money overall as in America, the yearly cost of treating PCOS is $4.36 billion.

ELIGIBILITY:
Inclusion Criteria:

* Women with PCOS

Exclusion Criteria:

* use of complimentary therapies within 6/12 prior to recruitment
* BMI >35
* taken combined oral contraceptives, metformin, or cyclical progestogens within 3/12 prior to recruitment

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-12; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To identify the most appropriate primary outcome measure for the ensuing RCT | Week 30

SECONDARY OUTCOMES:
Attainment of normal menstrual cycle length (i.e. 21-35 days) | 1 (baseline), week 10 (end of treatment) and week 30 (end of study)
Hormonal imbalances and irregular menses (commonly regarded at 6 cycles per annum or less) | 1 (baseline), week 10 (end of treatment) and week 30 (end of study)
weight, body mass index (BMI), hirsutism, thinning hair | week 1 (baseline), week 10 (end of treatment) and week 30 (end of study)
Fasting Insulin and blood sugar levels | week 1 (baseline), week 10 (end of treatment) and week 30 (end of study)
Quality of Life | week 1 (baseline), week 10 (end of treatment) and week 30 (end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn-Marie Walker, PhD, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham Hospitals, Nottingham, Nottingham, United Kingdom